CLINICAL TRIAL: NCT02112708
Title: Evaluation of the Effectiveness of Rational Emotive Behavioral Therapy (REBT/CBT) as an Intervention Tool in Clinical Social Work Consultation to Primary Care.
Brief Title: Cognitive Behavioral Therapy (REBT/CBT) Evaluation for Dysthymia in the Practice of Clinical Social Work at Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P13/035
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2014-03

CONDITIONS: Depression; Dysthymia; Ambulatory Health Services
Keywords: Psychotherapy, Rational-Emotive; Depression; Social Work; Primary Health Care
MeSH Terms: conditions — Depression; Dysthymic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rational-Emotive-Behavioral Therapy (Experimental): A social worker held eight 30 minutes sessions fortnightly of Rational-Emotive-Behavioral Therapy. First session is informative about the type of treatment to be performed. The next sessions work events, thoughts and feelings with the goal of changing the dysfunctional thoughts by other more rational ones, measured by scales.
  Interventions: Other: Rational-Emotive-Behavioral Therapy
- Control Group (Active Comparator): The control group (GC) will take the usual medical care for dysthymia, according with up-dated guidelines.
  Interventions: Other: Control Group usual care

INTERVENTIONS:
Other: Rational-Emotive-Behavioral Therapy — A social worker held eight 30 minutes sessions fortnightly. First session is informative about the type of treatment to be performed. The next sessions work events, thoughts and feelings with the goal of changing the dysfunctional thoughts by other more rational ones, measured by scales.
  Other Names: Cognitive-Emotive-Behavioral Therapy; REBT; CBT; REBT-CBT
  Arms: Rational-Emotive-Behavioral Therapy
Other: Control Group usual care — In the control group the dysthymia is treated as usual with the conventional treatment.
  Other Names: conventional treatment; usual care
  Arms: Control Group

SUMMARY:
Introduction: Minor psychiatric disorders are important in primary care, because of its high prevalence and consumption of healthcare resources generated.

Objective: Evaluate the effectiveness of rational emotive behavioral therapy (REBT), as an instrument of social work intervention to enhance changes in the parameters of quality of life, medical consultations and drug use in patients with dysthymia.

Design: Multicenter, prospective, not randomized clinical trial, with intervention and control group simultaneously in urban primary care settings and 1 year of follow up.

Participants: Out-patients seen in two Primary Care centers diagnosed with dysthymia according to DSM-IV classification of American Psychiatric Association.

Intervention: Subjects receive up to 8 biweekly individual sessions of thirty minutes of REBT administered by the Social Worker.

Variables: Demographic data, educational level, coexistence, comorbidity, quality of life assessment, severity of depression, number of visits to the General Practitioner (GP) and drug consumption: sedatives / antidepressants.

Expected Results: The expected results of the intervention, estimated from previous data, are:

* A decrease in attendance at medical visits per year
* An improvement in perceived quality of life, measured as values of the Quality of Life (QOL) questionnaire (Baker & Intagliata)
* An improvement in severity of depression, measured according to the Beck Depression Inventory.
* A reduction of treatment with psychotropic drugs (sedatives and antidepressants).

Potential impact expected: The investigators hope that rational emotive theory is an effective intervention method for handling minor psychiatric disorders in clinical social work.

DETAILED DESCRIPTION:
The calculation of the size of the population sample was performed for the worst case comparison of different outcome variables, so for a final ratio of 8% people taking hypnotics in Intervention Group (IG) versus 37% in the Control Group (CG), with significance level of 5% and a statistical power of 80%, previewing a 20% loss to follow-up and a ratio of 1 control per case, we need 50 individuals in the CG and 50 individuals in the IG.

Regarding to the attendance to primary care centers, was categorized as "improved" and "not improved or remains the same." "Improvement" is when the number of visits decrease over the previous year, comparing baseline data with respect 12 months. Also, improvement in the use of psychotropic medication is when intakes fall in the previous year by comparing baseline data with respect 12 months. When no data were available at 12 months, the comparison was made with data collected at 4 months.

Patients in IG were recruited from primary care center Sant Andreu, while the CG were enrolled in the primary care center in Martorell. The selection of the two groups in separate centers was determined to avoid the possible effects of contamination bias of the CBT-REBT. In the IG, each physician systematically derived patients with inclusion criteria to the social worker. In the CG, the physician made ordinary care task. In both groups, the number of visits to primary care centers and consumption of psychotropic drugs were extracted from the medical record and other information was obtained through interviews at baseline, 4 and 12 months.

All patients signed informed consent at baseline. In order to recruit homogeneous cases, clearly diagnosed and ensure comparability training for all recruiters was conducted. Collection forms and the database did not include confidential information to ensure confidentiality and anonymity, keeping a separately single list with relation to the number of each case.

Access data base was used to systematize the registration data collection and handling errors by different professionals. Previous comparison of baseline data between completers and dropouts, as well as between the IG and CG was performed by Chi-square and mean comparison. A descriptive analysis of baseline variables as frequencies, means, and dispersion measures was carried out. For the analysis of post-intervention improvement in outcome parameters in one group compared with another, only data from the baseline and 12 months were taken into account. Bivariate and multivariate analysis was performed using logistic regression to control for confounding factors. Values less than 0.05 were considered significant. The Statistical Package for the Social Sciences (SPSS) v.18 software was used.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis fo dysthymia
* Aged 14 or older

Exclusion Criteria:

* Impaired cognitive ability
* Illiteracy
* Refuses treatment
* Severe psychiatric disorders
* Participation in psychoeducational groups or other similar therapies.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carme Rovira Aler, LCSW, Principal Investigator — Catalan Institute of Health
Locations (1):
- Catalan Health Institute. ABS Sant Andreu 9D, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non randomized assignment: patients from Barcelona were assigned to Intervention Group and Patients from Martorell , assigned to Control Group.
Groups:
- Intervention Group: The intervention group received REBT by the purposely trained Social Worker at Barcelona
- Control Group: the control group received the standard medical care by their General Practitioner (GP) at Martorell
Period: Baseline
Arm/Group | Intervention Group | Control Group
Started | 79 | 50
Completed | 51 | 39
Not Completed | 28 | 11
Not completed — Physician Decision | 16 | 11
Not completed — Lost to Follow-up | 12 | 0
Period: 4 Month
Arm/Group | Intervention Group | Control Group
Started | 51 | 39
Completed | 39 | 38
Not Completed | 12 | 1
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 12 | 0
Period: 12 Month
Arm/Group | Intervention Group | Control Group
Started | 39 | 38
Completed | 39 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 51 | 39 | 90
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, continuous (years) | 60.8 (11.5) | 65.5 (13.2) | 62.86 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 34 | 83
  Male | 2 | 5 | 7
Educational level [Count of Participants; unit: Participants]
  Primary schooling | 27 | 32 | 59
  Secondary schooling and University | 24 | 7 | 31
Living arrangements [Count of Participants; unit: Participants]
  Lives on his/her own | 14 | 5 | 19
  Lives with other people | 37 | 32 | 69
psychopharmacological agents [Count of Participants; unit: Participants] — This measure take in account if participant takes or not psychopharmacological agents
  Participants
    No treatment | 6 | 4 | 10
    treatment | 45 | 35 | 80
Sedative-hypnotics agents [Count of Participants; unit: Participants]
  no | 44 | 28 | 72
  yes | 7 | 11 | 18
Antidepressants agents [Count of Participants; unit: Participants]
  no | 8 | 7 | 15
  yes | 43 | 32 | 75
Anxiolytic agents [Count of Participants; unit: Participants]
  no | 28 | 17 | 45
  yes | 23 | 22 | 45
Number of visits [Mean (Standard Deviation); unit: visits] — Number of visits to GP during previous year
  visits | 4 (2.9) | 2.2 (2.7) | 3.2 (2.95)
Number of psycopharmacological agents [Mean (Standard Deviation); unit: agents] — Number of psycopharmacological agents at baseline
  agents | 1.4 (0.8) | 1.7 (0.9) | 1.53 (.82)
Beck depression inventory score at baseline [Mean (Standard Deviation); unit: scores on a scale] — The Beck Depression Inventory is used in the detection and quantification of depressive symptoms in patients.
  It is a paper and pencil self-report made up of 21 Likert-type items. Its items are not derived from any specific theory about the construct measured, but instead describe the most frequent clinical symptoms of psychiatric patients with depression.
  Cut-off points have been established:
  [0-9: no depression], [10-18: mild depression], [19-29: moderate depression], [≥30: severe depression] The minimum and maximum scores on the scale are 0 and 63.
  scores on a scale | 24.5 (9.9) | 22.2 (11.7) | 23.50 (10.70)
Number of comorbidities [Mean (Standard Deviation); unit: comorbidities] — Number of comorbidities at baseline
  comorbidities | 2.9 (1.2) | 4.3 (2.1) | 3.47 (1.78)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Severity of Depression, Measured According to the Beck Depression Inventory, at 4 and 12 Months.
Description: The Beck Depression Inventory (BDI) consisted of twenty-one questions about how the subject has been feeling in the last week. Each question has a set of at least four possible answer choices, ranging in intensity.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-offs are as follows:
  * 0-9: indicates minimal depression
  * 10-18: indicates mild depression
  * 19-29: indicates moderate depression
  * 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
Time Frame: Baseline, month 4, month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 51 | 38
score on a scale
  12 months analysis | 16.18 (11.50) | 19.90 (14.43)
  4 months analysis | 16.29 (10.50) | 20.90 (13.70)
  Baseline analysis | 24.5 (9.9) | 22.2 (11.7)

2. Secondary Outcome: Change From Baseline in Perceived Quality of Life, Measured as Values of Satisfaction With Life Domains Scale (SLDS) at 4 and 12 Months
Description: The Satisfaction with Life Domains Scale (SLDS) is a measure of respondent satisfaction constructed to assess patient's satisfaction regarding 15 life domains.
  The respondent is asked in each of 15 domains to indicate his/her feelings by choosing one of seven faces ranging from a "delighted" face with a large upturned smile (scored 7) to a "terrible" face with a deep frown (scored 1).
  The patients are asked to pick the face that best represented their degree of satisfaction with the proposed life areas.
  The last of the life areas (The place they live in currently compared with the state hospital) has been discarded for our study, because the patients were treated by primary care.
  The overall scale (summatory of 15 domains) runs from minimum as 0 to maximum as 98
Time Frame: Baseline, month 4, month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 51 | 38
score on a scale
  12 months analysis | 5.02 (1.48) | 4.59 (1.39)
  4 months analysis | 5.00 (1.01) | 4.60 (1.50)
  Baseline analysis | 4.43 (1.01) | 4.60 (1.24)

3. Other Pre Specified Outcome: Average Number of Visits of Attendance at Medical Visits in Previous Year and 1 Year of Follow up Date.
Description: Attendance means at medical visits were obtained from computerized medical records for a period of one year previous to the baseline date and 1 year of follow up date.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: medical visits attended
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 51 | 38
medical visits attended
  Baseline | 4.0 (2.9) | 2.2 (2.7)
  1 year of follow up date | 1.4 (1.7) | 1.7 (2.3)

4. Other Pre Specified Outcome: Percentage of People in the Group Who Stop Taking or Reduce the Dose of Psychotropic Drugs at 12 Months
Description: Percentage of people with any improvement in the dosage of psychotropic drugs (sedatives and antidepressants) in the group at 12 months compared to the baseline date of the study.
Time Frame: Baseline, months 12
Measure: Number (95% Confidence Interval); unit: Percentatge of people with any improveme
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 51 | 38
Percentatge of people with any improveme | 47.8 [34.8 to 61.2] | 11.4 [4.7 to 25.2]

ADVERSE EVENTS:
Time Frame: 1 year
Description: The occurrence of death due to any cause is the only adverse event reported because this is a psychosocial intervention.
Arm/Group | Rational-Emotive-Behavioral Therapy | Control Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/39
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/39
Other Adverse Events (participants affected / at risk) | 0/51 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No